CLINICAL TRIAL: NCT00270335
Title: Optimizing Propofol in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Lars S. Rasmussen, Department of Anaesthesia, HOC, Copenhagen University Hospital, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-005400-17; GCP-2005-087; KF 02 284302
Record Dates: First submitted 2005-12-23; First posted 2005-12-26 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): General anesthesia titrated according to a cerebral state monitor
  Interventions: Drug: Propofol
- B (Active Comparator): General anesthesia titrated according to usual clinical criteria
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol

SUMMARY:
An accurate dosage of anesthetics during surgery is important. Usually this is achieved through close observation of the patient, but a new monitor (CSM-monitor) can measure the level of anesthesia more closely.

In obese patients dosage of drugs is difficult due to the change in body composition. The CSM-monitor may provide a more accurate dosage of propofol (an anesthetic agent) during surgery, and as a consequence of that, also reduce the postoperative need for analgesics.

Main objective: To optimise propofol dosing in obese patients undergoing hysterectomy.

Main hypothesis: Monitoring the depth of anesthesia using the CSM-monitor reduces time to opening eyes in obese patients after hysterectomy in propofol anesthesia.

Secondary hypotheses: CSM-monitoring reduce propofol dose in obese patients undergoing hysterectomy. Patients with a high CSM-level during hysterectomy have higher postoperative consumption of analgesics. Supplementary, an algorithm for the dose of propofol that most frequently results in a CSM-level between 40 and 60 is calculated.

ELIGIBILITY:
Inclusion Criteria:

* Elective abdominal non-laparoscopic hysterectomy
* Age > 18 years
* ASA physical status I-III
* Body Mass Index 30 or above

Exclusion Criteria:

* Allergic towards propofol
* Daily consumption of benzodiazepines (more than at nighttime), opioids or amphetamine preoperatively.
* Disease with expected EEG-abnormality or impaired auditory function: Epilepsy, deafness, previous neurosurgery, previous or actual neurologic disease with neurologic deficit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to opening eyes in obese patients after hysterectomy in propofol anaesthesia.

SECONDARY OUTCOMES:
Propofol dose in obese patients undergoing hysterectomy.
Postoperative consumption of analgesics. | 24 h after surgery
The algorithm for the dose of propofol that most frequently results in a CSM-level between 40 and 60.

CONTACTS AND LOCATIONS:
Overall Officials: Lars S. Rasmussen, MD, PhD, Study Chair — Department of anesthesia, 4231, Center of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet
Locations (2):
- Denmark (2):
  - Department of Anaesthesia, Juliane Marie Centre, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Department of Anaesthesia, Copenhagen University Hospital Herlev, Herlev

REFERENCES:
- [Result] Meyhoff CS, Henneberg SW, Jorgensen BG, Gatke MR, Rasmussen LS. Depth of anaesthesia monitoring in obese patients: a randomized study of propofol-remifentanil. Acta Anaesthesiol Scand. 2009 Mar;53(3):369-75. doi: 10.1111/j.1399-6576.2008.01872.x. Epub 2009 Jan 23. PMID 19173688